CLINICAL TRIAL: NCT00127660
Title: Effect of Nutrition Labeling on Fast Food Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: DK67599 (completed); R01DK067599 (NIH)
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Menu: calories=yes, value pricing=no (Experimental): There were calories listed on the menu, but no value pricing was in place.
  Interventions: Behavioral: Menu: calories=yes, value pricing=no
- Menu: calories=yes, value pricing = yes (Experimental): There were calories listed on the menu, AND value pricing was in place.
  Interventions: Behavioral: Menu: calories=yes, value pricing = yes
- Menu: calories=no, value pricing = no (Experimental): Calories were not listed on the menu, and value pricing was not in place.
  Interventions: Behavioral: Menu: calories=no, value pricing = no
- Menu: calories=no, value pricing = yes (No Intervention): CONTROL CONDITION: calories were not listed on the menu, and value pricing WAS in place.

INTERVENTIONS:
Behavioral: Menu: calories=yes, value pricing=no
  Arms: Menu: calories=yes, value pricing=no
Behavioral: Menu: calories=yes, value pricing = yes
  Arms: Menu: calories=yes, value pricing = yes
Behavioral: Menu: calories=no, value pricing = no
  Arms: Menu: calories=no, value pricing = no

SUMMARY:
A study examining menu choices made at fast food restaurants.

DETAILED DESCRIPTION:
To examine the effect of point-of-purchase calorie information and value size pricing on fast food meal choices a randomized 2 × 2 factorial experiment was conducted in which participants ordered a fast food meal from one of four menus that varied with respect to whether calorie information was provided and whether value size pricing was used.

ELIGIBILITY:
Inclusion Criteria:

* Must be 16 years old or older
* Must regularly eat at fast food restaurants

Exclusion Criteria:

* Non-english speakers

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Harnack, DrPH, Principal Investigator — University of Minnesota
Locations (1):
- Division of Epidemiology & Community Health, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Harnack LJ, French SA, Oakes JM, Story MT, Jeffery RW, Rydell SA. Effects of calorie labeling and value size pricing on fast food meal choices: results from an experimental trial. Int J Behav Nutr Phys Act. 2008 Dec 5;5:63. doi: 10.1186/1479-5868-5-63. PMID 19061510
- [Result] Fitch RC, Harnack LJ, Neumark-Sztainer DR, Story MT, French SA, Oakes JM, Rydell SA. Providing calorie information on fast-food restaurant menu boards: consumer views. Am J Health Promot. 2009 Nov-Dec;24(2):129-32. doi: 10.4278/ajhp.08031426. PMID 19928485
- [Result] Rydell SA, Harnack LJ, Oakes JM, Story M, Jeffery RW, French SA. Why eat at fast-food restaurants: reported reasons among frequent consumers. J Am Diet Assoc. 2008 Dec;108(12):2066-70. doi: 10.1016/j.jada.2008.09.008. PMID 19027410

RESULTS

PARTICIPANT FLOW:
Groups:
- Menu: Calories=Yes, Value Pricing=no: Calories listed on menu, but value pricing was not in place.
- Menu: Calories=Yes, Value Pricing = Yes: Calories listed on menu, value pricing in place.
- Menu: Calories=no, Value Pricing = no: Calories not listed on menu, value pricing not in place
- Menu: Calories=no, Value Pricing = Yes: CONTROL CONDITION: calories not listed on menu, value pricing in place.
Period: Overall Study
Arm/Group | Menu: Calories=Yes, Value Pricing=no | Menu: Calories=Yes, Value Pricing = Yes | Menu: Calories=no, Value Pricing = no | Menu: Calories=no, Value Pricing = Yes
Started | 153 | 154 | 148 | 150
Completed | 150 | 151 | 143 | 150
Not Completed | 3 | 3 | 5 | 0
Not completed — Protocol Violation | 3 | 3 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menu: Calories=Yes, Value Pricing=no | Menu: Calories=Yes, Value Pricing = Yes | Menu: Calories=no, Value Pricing = no | Menu: Calories=no, Value Pricing = Yes | Total
Number analyzed (Participants) | 150 | 151 | 143 | 150 | 594
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 30 | 45 | 40 | 147
  Between 18 and 65 years | 95 | 92 | 80 | 96 | 363
  >=65 years | 23 | 29 | 18 | 14 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 94 | 89 | 89 | 353
  Male | 69 | 57 | 54 | 61 | 241
Region of Enrollment [Number; unit: participants]
  United States | 150 | 151 | 143 | 150 | 594

OUTCOME MEASURES:

1. Primary Outcome: Total Calories of Meal Ordered
Time Frame: single study visit
Reporting Status: Not Posted

2. Primary Outcome: Energy Intake
Description: energy content of meal ordered and consumed.
Time Frame: After meal
Measure: Mean (Standard Deviation); unit: kcal/meal
Arm/Group | Menu: Calories=Yes, Value Pricing=no | Menu: Calories=Yes, Value Pricing = Yes | Menu: Calories=no, Value Pricing = no | Menu: Calories=no, Value Pricing = Yes
Number analyzed (Participants) | 150 | 151 | 143 | 150
kcal/meal | 842.3 (425.3) | 873.6 (439.1) | 881.7 (353.6) | 827.5 (400.6)

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | Menu: Calories=Yes, Value Pricing=no | Menu: Calories=Yes, Value Pricing = Yes | Menu: Calories=no, Value Pricing = no | Menu: Calories=no, Value Pricing = Yes
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Meal choices were tested on just one occasion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No